CLINICAL TRIAL: NCT00608075
Title: Neurofunctional and Neurochemical Markers of Treatment Response in Bipolar Disorder
Acronym: LAMBS/LADS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Caleb M. Adler, Associate Professor, University of Cincinnati
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Adler #1; R01-0788043-01A1
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Manic Patients
  Interventions: Drug: lithium
- 2 (Other): Depressed Patients
  Interventions: Drug: Lithium

INTERVENTIONS:
Drug: lithium — 600 mg - 1800 mg per day
  Arms: 1
Drug: Lithium — 600 - 1800 mg
  Arms: 2

SUMMARY:
The purpose of the research is to study brain structure, function and chemistry of patients with bipolar disorder who are receiving lithium, an FDA-approved treatment for bipolar mania, in order to better understand who benefits from treatment and why they respond to medications. Studying this may help improve treatment and outcome in patients with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria- bipolar patients (Manic=, depressed=60; 30 patients/year):

1. The patient meets DSM-IV criteria for type I bipolar disorder, manic or mixed, or depressed.
2. The patient has an index Young Mania Rating Scale (YMRS)total score >15 or Montgomery Asberg Rating Scale (MADRS) total score >20.
3. The patient is between 15 and 55 years old.

Inclusion Criteria- Healthy subjects (N=40):

1. Healthy subjects will be between the ages of 15 and 55 years.
2. Healthy subjects will have no history of any Axis I psychiatric disorder.
3. Healthy subjects will have no first-degree relatives with affective or psychotic disorders.

Exclusion criteria: All subjects will be excluded from participation for the following reasons.

1. Any medical or neurological disorder that could influence fMRI and MRS results.
2. A history of mental retardation or an estimated IQ total score <85.
3. An MRI scan is contraindicated in the subject for any reason, including psychological impediments to being inside the MR scanner.
4. The patient cannot attend follow-up visits.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 260 (Estimated)
Dates: Start 2007-04; Primary Completion 2015-07 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The purpose of the research is to study brain structure, function and chemistry of patients with bipolar disorder who are receiving lithium. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Caleb M Adler, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Lei D, Li W, Tallman MJ, Strakowski SM, DelBello MP, Rodrigo Patino L, Fleck DE, Lui S, Gong Q, Sweeney JA, Strawn JR, Nery FG, Welge JA, Rummelhoff E, Adler CM. Changes in the structural brain connectome over the course of a nonrandomized clinical trial for acute mania. Neuropsychopharmacology. 2022 Oct;47(11):1961-1968. doi: 10.1038/s41386-022-01328-y. Epub 2022 May 18. PMID 35585125